CLINICAL TRIAL: NCT06243627
Title: A Single-Center, Comparative, Randomized, Safety-in-Use Clinical Study to Assess Skin Acceptability and Efficacy in Improving Skin Barrier Function of Two Facial Sunscreens in Adult Participants With Sensitive Skin
Brief Title: A Study to Assess Safety and Improvement in Skin Barrier After Using 2 Facial Sunscreens in Adults With Sensitive Skin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Consumer Inc. (J&JCI) (Industry)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CCSSKA005438
Record Dates: First submitted 2024-01-29; First posted 2024-02-06 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-01

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arm 1: Sunscreen C Color 2.0 Sun Protection Factor (SPF) 70 and Sunscreen M Very Light SPF 50 (Experimental): The participants will apply topically two colored sunscreens: C color 2.0 and M very light, one on each half of the face at least twice a day for 21 days.
  Interventions: Other: Sunscreen C Color 2.0 SPF 70; Other: Sunscreen M Very Light SPF 50
- Arm 2: Sunscreen C Color 2.0 SPF 70 and Sunscreen M Golden Color SPF 50 (Experimental): The participants will apply topically two colored sunscreens: C color 2.0 and M golden color, one on each half of the face at least twice a day for 21 days.
  Interventions: Other: Sunscreen C Color 2.0 SPF 70; Other: Sunscreen M Golden Color SPF 50
- Arm 3: Sunscreen C Color 3.0 SPF 70 and Sunscreen M Very Light SPF 50 (Experimental): The participants will apply topically two colored sunscreens: C color 3.0 and M very light, one on each half of the face at least twice a day for 21 days.
  Interventions: Other: Sunscreen C Color 3.0 SPF 70; Other: Sunscreen M Very Light SPF 50
- Arm 4: Sunscreen C Color 3.0 SPF 70 and Sunscreen M Golden Color SPF 50 (Experimental): The participants will apply topically two colored sunscreens: C color 3.0 and M golden color, one on each half of the face at least twice a day for 21 days.
  Interventions: Other: Sunscreen C Color 3.0 SPF 70; Other: Sunscreen M Golden Color SPF 50

INTERVENTIONS:
Other: Sunscreen C Color 2.0 SPF 70 — Sunscreen C color 2.0 SPF 70 will be applied topically on half of the face.
  Other Names: E003431A-01
  Arms: Arm 1: Sunscreen C Color 2.0 Sun Protection Factor (SPF) 70 and Sunscreen M Very Light SPF 50; Arm 2: Sunscreen C Color 2.0 SPF 70 and Sunscreen M Golden Color SPF 50
Other: Sunscreen C Color 3.0 SPF 70 — Sunscreen C color 3.0 SPF 70 will be applied topically on half of the face.
  Other Names: E003431A-02
  Arms: Arm 3: Sunscreen C Color 3.0 SPF 70 and Sunscreen M Very Light SPF 50; Arm 4: Sunscreen C Color 3.0 SPF 70 and Sunscreen M Golden Color SPF 50
Other: Sunscreen M Very Light SPF 50 — Sunscreen M very light SPF 50 will be applied topically on half of the face.
  Other Names: E003431A-03
  Arms: Arm 1: Sunscreen C Color 2.0 Sun Protection Factor (SPF) 70 and Sunscreen M Very Light SPF 50; Arm 3: Sunscreen C Color 3.0 SPF 70 and Sunscreen M Very Light SPF 50
Other: Sunscreen M Golden Color SPF 50 — Sunscreen M golden color SPF 50 will be applied topically on half of the face.
  Other Names: E003431A-04
  Arms: Arm 2: Sunscreen C Color 2.0 SPF 70 and Sunscreen M Golden Color SPF 50; Arm 4: Sunscreen C Color 3.0 SPF 70 and Sunscreen M Golden Color SPF 50

SUMMARY:
The purpose of this trial is to evaluate 1) the dermatological tolerability of 2 facial sunscreens after 21 (+2) days of use under normal conditions on the half face by adult subjects with sensitive skin, 2) Compare the efficacy of investigational products (IPs) after 21 (+2) days of use in adult subjects with sensitive skin, under dermatological supervision through the following evaluations: the transepidermal water loss in the nasolabial region; the sensory perception of the subjects using the sensory perception questionnaire, after 21 (+2) days of use under normal conditions; the sensitivity of the subjects' skin after the first application of each product using a questionnaire on the perception of signs of discomfort.

ELIGIBILITY:
Inclusion Criteria:

* Participants vaccinated against coronavirus disease 2019 (COVID-19)
* Participants of any gender
* Participants of any ethnicities according to Brazilian Institute of Geography and Statistics (IBGE) criteria
* Phototype II to IV according to Fitzpatrick's classification
* Participants - in good health based on medical history reported by the subject
* Participants presenting intact skin on the face, with the exception of clinical signs characteristic of sensitive skin
* Participants who declare themselves as having sensitive skin (according to the Institute's sensitive skin questionnaire, completed in the recruitment phase and reconfirmed by the physician on the day of inclusion)
* Able to read, write, speak and understand Portuguese (able to read and understand the documents delivered and what is explained to them)
* Participants who agree to maintain their cosmetic habits during the study period
* Participants who agree to maintain their cosmetic habits during the study period
* Participant who signed the Informed Consent Document (ICD)
* Agreement to adhere to the procedures and requirements of the study and to attend the Site on the day(s) and time(s) determined for the assessments
* Participant that intend to complete the study and is willing and able to follow all study instructions

Exclusion Criteria:

* Participants that have had allergies or adverse reactions to common topical skincare products, including sunscreens, medications, or other products that the investigator considers relevant
* Participants that present a skin condition that may influence the study results (specifically psoriasis, eczema, atopic dermatitis, cutaneous xerosis, intense erythema, or active skin cancer). Mild erythema and xerosis associated with a sensitive skin condition are acceptable for eligibility
* Participants that present primary/secondary lesions (for example: scars, ulcers, vesicles, vitiligo) or tattoos on the test areas
* Participants that have undertaken cosmetic or dermatological treatment, invasive or non-invasive, in the test areas within 3 weeks before the beginning of the study and during the study
* Participants that have self-reported Type 1 or Type 2 diabetes or are taking insulin or another anti-diabetic medication
* Participants that are taking a medication that would mask an adverse event (AE) or influence the study results, including: Immunosuppressive or steroidal drugs within 2 months before Visit 1; Non-steroidal anti-inflammatory drugs within 5 days before Visit 1; Antihistamines within 2 weeks before Visit 1. If an individual is taking one of these medication types, the individual is not considered eligible at screening. However, if a subject begins using one of these medications during the study, the study physician should be consulted to consider the impact of the specific medication on subject safety and/or the study results, as described in section "Concurrent/Concomitant Medication"
* Participants that are self-reported to be pregnant or planning to become pregnant during the study
* Participants that have a history of a health condition/situation which may put the individual at significant risk, influence the study results, or interfere significantly with the individual's participation in the study
* Participants that are simultaneously participating in any other study
* Participants that are employees/contractors or immediate family members of the principal investigator (PI), study site, or sponsor
* History of non-adherence or unwillingness to adhere to the study protocol
* Any condition not previously mentioned that, in the opinion of the PI, may compromise the study evaluation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2023-09-27 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-12-11 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in Dermatological Tolerability | Baseline (Day 1), Day 21
  Change from baseline in dermatological tolerability will be reported. Dermatological tolerability includes a clinical assessment of the participant's initial skin condition, carried out by the study dermatologist according to the Skin Reaction Intensity Assessment Scale. Skin reaction intensity assessment of erythema, edema, blistering and peeling on the face will be done. Each skin reaction was scored on 4-point scale 0 = absent, 1 = mild, 2 =moderate, and 3 = intense. A decrease in score at post-baseline timepoints compared to baseline indicates an improvement.
Change From Baseline in Skin Barrier Integrity | Baseline (Day 1), Day 21
  Change from baseline in skin barrier integrity will be reported. The facial skin barrier will be assessed by a trained technician using instrumental measurements with the Tewameter TM 300. The Tewameter measures transepidermal water loss (TEWL) that is the flow of water out of the skin. TEWL measurement will be taken in the nasolabial region of each half of the face.
Number of Participants With Sensory Perception as Assessed by Sensory Perception Questionnaire | At Day 21
  Number of participants with sensory perception as assessed by sensory perception questionnaire will be reported. The sensory perception of each sunscreen will be concluded from the data obtained from the sensory perception questionnaire which includes overall satisfaction, skin and eye irritation, comfort and other characteristics (stickiness, lightness etcetera). Sensory perception questionnaire includes 1 question on overall satisfaction with sunscreen by scoring on a scale ranged from 1 to 7, 1= disliked very much and 7= liked very much; 3 questions with participant's response on "does not irritate the skin, eye and felt comfortable using the sunscreen" on a response scale ranging from 1 to 5, 1= strongly disagree and 5= strongly agree; and 1 question that correlate the characteristic (stickiness, lightness etcetera.) with each product tested.
Number of Participants With Skin Sensitivity as Assessed by Discomfort Questionnaire | At Day 1
  Number of participants with skin sensitivity as assessed by perception questionnaire on discomfort signs will be reported. Assessment of skin sensitivity after application of each sunscreen will be concluded from the data obtained by filling in the questionnaire on the perception of signs of discomfort. Perception questionnaire on discomfort signs includes sensation of discomfort, burning sensation, itching, redness sensation on skin and eye irritation. For each sign the participant will select a response on a scale ranging from 0 to 9, where 0 = no discomfort sign and 9= intense discomfort sign. Higher score indicates intense discomfort sign. If a participant has a moderate or/to intense reaction (from 4 to 9) an adverse event will be open.
Number of Participants With Adverse Events | Up to Day 21
  Number of participants with adverse events will be reported. An adverse event is any untoward medical occurrence in a clinical study participant temporally associated with the clinical investigation, whether or not the event has a causal relationship to the participants' participation in the trial. It is therefore any unfavorable and unintended sign (including an abnormal finding), symptom, or disease that occurs during the trial. This can include any occurrence that is new in onset, an aggravation of severity/frequency of a baseline condition, or abnormal results of diagnostic procedures, including laboratory test abnormalities.

CONTACTS AND LOCATIONS:
Overall Officials: Gabrielli Brianezi, Principal Investigator — Johnson & Johnson Consumer Inc. (J&JCI)
Locations (1):
- Allergisa Pesquisa Dermato-Cosmetica Ltda, Campinas, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Consumer Inc. has an agreement with the Yale Open Data Access (YODA) Project to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu.
URL: http://yoda.yale.edu.